CLINICAL TRIAL: NCT03855709
Title: Patterns of Antibiotic Resistant Bacterial Infections in Liver Intensive Care Unit
Brief Title: Antibiotic-resistant Bacterial Infection of Hepatic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karema Azoz Mostafa, Specialist, Assiut University
Other Study IDs: bacterial resistence
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Antibiotic Resistant Infection; Liver Cirrhoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: microbiological culture and sensetivity — microbioloical culture will be used to detect microbiological profile in hepatic patients with infections, drug sensitivity to detect resistent bacteria which will be confirmed using PCR detection of resistent gene

SUMMARY:
the investigators want to identify the microbial profile, antibiotic resistant bacteria in hepatic patients with infections in Liver ICU, and explore risk factors and outcomes in those patients with antibiotic resistant bacteria.

DETAILED DESCRIPTION:
Bacterial infection signifies major clinical challenge in cirrhotic patients where about 35% of these patients acquire hospital-acquired infections compared with 5% of other hospital in-patients without cirrhosis.It is associated with a mortality rate of 38% with a four-fold increase compared to individuals without cirrhosis.

Cirrhotic patients have a high risk for antimicrobial resistance because of chronic use of prescribed antibiotics like quinolones in secondary prophylaxis for spontaneous bacterial peritonitis. In addition, undergoing invasive procedures and recurrent hospital admissions encourage both increased occurrence of antimicrobial resistance and the spread of resistant pathogens in these patients.

Epidemiology, risk factors and clinical outcomes of MDR infections have raised a special attention in cirrhosis. Some studies reported bacterial resistance in about 50% of examined patients and it is associated with treatment failure, septic shock and hospital mortality especially in nosocomial and healthcare related infections

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESLD at Liver ICU. All patients have the diagnostic criteria for liver cirrhosis by clinical, biochemical, and ultrasonography findings. The severity of liver cirrhosis will be assessed according to the Child-Pugh classification and model for end-stage liver disease (MELD) score.
* These patients are diagnosed as having infection at admission or acquire infection during hospitalization.

Exclusion Criteria:

* Age ≤ 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed to have ESLD admitted to EL-Rajhi liver hsopital (Assiut university hopsitals) diagnosed to have infection at admission or develop infection during hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Detection of different bacterial causing infections in hepatic patients | baseline
  Bacteriological cultures will be performed with VITEK 2 COMPACT-15 automated system (bioMerieux Inc, Mercy L'etoil, Fransa).
To detect antibiotic resistant bacteria among these patients. | baseline
  molecular detection of genes responsible for antibiotic resistance using PCR for isolates bacteria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez J, Acevedo J, Castro M, Garcia O, de Lope CR, Roca D, Pavesi M, Sola E, Moreira L, Silva A, Seva-Pereira T, Corradi F, Mensa J, Gines P, Arroyo V. Prevalence and risk factors of infections by multiresistant bacteria in cirrhosis: a prospective study. Hepatology. 2012 May;55(5):1551-61. doi: 10.1002/hep.25532. Epub 2012 Apr 4. PMID 22183941
- [Background] Fernandez J, Navasa M, Gomez J, Colmenero J, Vila J, Arroyo V, Rodes J. Bacterial infections in cirrhosis: epidemiological changes with invasive procedures and norfloxacin prophylaxis. Hepatology. 2002 Jan;35(1):140-8. doi: 10.1053/jhep.2002.30082. PMID 11786970
- [Background] Arvaniti V, D'Amico G, Fede G, Manousou P, Tsochatzis E, Pleguezuelo M, Burroughs AK. Infections in patients with cirrhosis increase mortality four-fold and should be used in determining prognosis. Gastroenterology. 2010 Oct;139(4):1246-56, 1256.e1-5. doi: 10.1053/j.gastro.2010.06.019. Epub 2010 Jun 14. PMID 20558165
- [Background] Merli M, Lucidi C, Di Gregorio V, Falcone M, Giannelli V, Lattanzi B, Giusto M, Ceccarelli G, Farcomeni A, Riggio O, Venditti M. The spread of multi drug resistant infections is leading to an increase in the empirical antibiotic treatment failure in cirrhosis: a prospective survey. PLoS One. 2015 May 21;10(5):e0127448. doi: 10.1371/journal.pone.0127448. eCollection 2015. PMID 25996499
- [Background] Merli M, Lucidi C. Bacterial resistance in cirrhotic patients: an emerging reality. J Hepatol. 2012 Apr;56(4):756-7. doi: 10.1016/j.jhep.2011.12.004. Epub 2012 Jan 8. No abstract available. PMID 22230869
- [Background] Shallcross L, O'Brien A. Antimicrobial resistance in liver disease: better diagnostics are needed. Lancet Gastroenterol Hepatol. 2017 Mar;2(3):151-153. doi: 10.1016/S2468-1253(16)30240-0. Epub 2017 Feb 9. No abstract available. PMID 28404125